CLINICAL TRIAL: NCT00462696
Title: Study Evaluating the Contribution of MRI for the Evaluation of Early Response to Neoadjuvant Chemotherapy in Patients With Infiltrative Breast Cancer
Brief Title: MRI in Evaluating Early Response to Chemotherapy in Women With Infiltrating Breast Cancer
Acronym: ISNA-Sein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IB-2005-37
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2025-09-15 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Woment treated with neoadjuvant chemotherapy for breast cancer (Experimental): The patient will be recruited during a multidisciplinary team meeting (MDT) involving a medical oncologist, radiation oncologist, and surgeon. The histological diagnosis of invasive breast cancer will be confirmed based on the results of the micro-biopsy, which will be performed during the MDT meeting, after the initial MRI scan. The patient will submit her signed informed consent form. The MRI will be performed before the micro-biopsy so as not to distort the measurement of the tumor volume by a possible post-collection hematoma.
  Interventions: Drug: Neoadjuvant chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy — Neoadjuvant tehrapy as per standard practice :
  Patients will be treated with six cycles of neoadjuvant chemotherapy combining epirubicin (75 mg/m² on day 1) and docetaxel (75 mg/m² on day 1), administered every 21 days (Delcambre, 2005; Wenzel, 1999). This treatment regimen is in line with the latest international recommendations (Kaufmann, 2003). The addition of a leukocyte growth factor in cases of grade IV leukopenia and/or treatment postponements due to grade 3-4 toxicity will be authorized with a maximum delay of 2 weeks per cycle. Dose reductions will be authorized in 25% increments for grade 3-4 toxicity
  . Systematic surgical excision of the residual lesion (or the initial tumor site) will be performed between 22 and 35 days after the last chemotherapy treatment, in the form of a lumpectomy or mastectomy, depending on the residual tumor. Lymph node dissection will be systematically associated.

SUMMARY:
RATIONALE: Diagnostic procedures, such as magnetic resonance imaging (MRI), may help in learning how well chemotherapy works to kill breast cancer cells and allow doctors to plan better treatment. Drugs used in chemotherapy, such as epirubicin and docetaxel, may stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This clinical trial is studying MRI in evaluating early response to chemotherapy in women receiving chemotherapy for infiltrating breast cancer.

DETAILED DESCRIPTION:
Pilot study (feasibility) without direct individual benefit aimed at breast cancer patients treated with neoadjuvant chemotherapy prior to local breast surgery (lumpectomy or mastectomy).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed infiltrative breast cancer meeting 1 of the following criteria:

  * Operable T2 or T3, M0 disease
  * Locally advanced disease (T4a, b, or c)

    * No T4d disease
* Indication for neoadjuvant chemotherapy before breast-conserving surgery

  * No desire by patient for complete mastectomy
* No overexpression of HER-2
* No multifocal tumor
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Life expectancy > 6 months
* No contraindication to MRI with contrast, including any of the following:

  * Claustrophobia
  * Prior major allergies
  * Cardiac pacemaker
  * Surgical clips
  * Certain cardiac valves
  * Sunken or hollow filters
  * Implanted pump
  * Cochlear implants
  * Metallic foreign body (intra-ocular)
* No contraindication to chemotherapy or surgery
* No other serious condition that would preclude study therapy
* No other uncontrolled medical condition, including any of the following:

  * Thyroid disease
  * Neuropsychiatric disease
  * Infection
  * Insufficient coronary capacity
  * NYHA class III-IV heart disease
* No HIV positivity
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy, radiotherapy, or surgery for ipsilateral breast cancer
* No prior biopsy of tumor before MRI
* No MRI at another center within the past 15 days
* No participation in another investigational study of anticancer therapy within the past 30 days

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2008-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Valentin, MD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Woment Treated With Neoadjuvant Chemotherapy for Breast Cancer: The patient will be recruited during a multidisciplinary team meeting (MDT). The histological diagnosis of invasive breast cancer will be confirmed based on the results of the micro-biopsy, which will be performed during the MDT meeting, after the initial MRI scan. The patient will submit her signed informed consent form. The MRI will be performed before the micro-biopsy so as not to distort the measurement of the tumor volume by a possible post-collection hematoma.
  Neoadjuvant chemotherapy: as per standard practice
Period: Overall Study
Arm/Group | Woment Treated With Neoadjuvant Chemotherapy for Breast Cancer
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Woment Treated With Neoadjuvant Chemotherapy for Breast Cancer
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 47 [38 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 16

OUTCOME MEASURES:

1. Primary Outcome: Reproducibility of the MRI Vascular Permeability (Kep)
Description: MRI vascular permeability is measured using Kep index (Rate constant between extracellular extravascular space (EES) and plasma).
  Kep index will be measured at the second cycle of neoadjuvant chemotherapy. MRI will be read independently by two radiologists experienced in breast imaging and breast MRI, blind to the results found by the other, in order to assess the reproducibility of the measurement.
Time Frame: two months after start of neoadjuvant chemotherapy
Population: Outcome could not be assessed. outcome was based on the assessment of MRI index by two radiologists. Only one radiologist assessed the index.
Arm/Group | Woment Treated With Neoadjuvant Chemotherapy for Breast Cancer
Number analyzed (Participants) | 0

2. Primary Outcome: Reproducibility of the MRI Vascular Permeability (HA)
Description: MRI vascular permeability is measured using HA index (Hepatic Artery index or Hepatic Arterial perfusion).
  HA index will be measured at the second cycle of neoadjuvant chemotherapy. MRI will be read independently by two radiologists experienced in breast imaging and breast MRI, blind to the results found by the other, in order to assess the reproducibility of the measurement.
Time Frame: two months after start of neoadjuvant chemotherapy
Population: as for outcome 1
Arm/Group | Woment Treated With Neoadjuvant Chemotherapy for Breast Cancer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Woment Treated With Neoadjuvant Chemotherapy for Breast Cancer
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes